CLINICAL TRIAL: NCT01647984
Title: Study on the Role of a Combination of Nutraceuticals (Ritmonutra) With an Effect on Benign Supraventricular and Ventricular Arrhythmias in Subjects Free of a Specific Organic Heart Disease.
Brief Title: Role of a Combination of Nutraceuticals (Ritmonutra) on Benign Supraventricular and Ventricular Arrhythmias
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruno Trimarco, Full Professor of Cardiology, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RITMONUTRA 2012
Record Dates: First submitted 2012-07-12; First posted 2012-07-24 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Ventricular and Atrial Extrasytoles
Keywords: Arrhythmias; Life quality
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Docosahexaenoic Acids; crataegus extract; astaxanthine; Vitamin E; Vitamin B Complex; Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Inert Placebo - Vitamin B complex + diet
  Interventions: Dietary Supplement: placebo
- Ritmonutra (Active Comparator): Omega-3 polyunsaturated fatty acids, Hawthorn, Astaxanthin, Vitamin E, Vitamin B complex + diet
  Interventions: Dietary Supplement: Ritmonutra

INTERVENTIONS:
Dietary Supplement: Ritmonutra — Ritmonutra ® contains: 720 mg of Fish Oil with Omega-3, including 480 mg of EPA and 40 mg of DHA, Hawthorn (extract from Crataegus mongyna) 300 mg equivalent to 5.4 mg of vitexin, 4 mg of Astaxanthin and 36 mg of Vitamin E
  Other Names: Omega-3 polyunsaturated fatty acids; Hawthorn; Astaxanthin; Vitamin E; Vitamin B complex; Diet
  Arms: Ritmonutra
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
Study on the role of a combination of nutraceuticals (Ritmonutra) with an effect on benign supraventricular and ventricular extrasystoles in subjects free of a specific organic heart disease. It has been suggested treatment with a nutritional supplement, able to normalize the 'cardiac electrophysiology' and help to maintain wellness. Ritmonutra ® is a combination of nutraceuticals®, including Omega-3 polyunsaturated fatty acids, Hawthorn, Astaxanthin and Vitamin E, help to normalize the heart pacing, reducing the total number of benign extrasystoles and consequently improving the quality of life.

DETAILED DESCRIPTION:
Benign supraventricular and ventricular extrasystoles may frequently occur in subjects free of a specific organic heart disease. use of potent anti-arrhythmic is not indicated for these kind of arrhythmias but the occurrence of this type of extrasystoles may generate concern in patients and consequently worse quality of life.

1. Study Rationale Supraventricular and ventricular extrasystoles may frequently occur in subjects free of a specific organic heart disease. The prognosis of these arrhythmias is benign and the only clinical indication is to perform periodic medical examinations to confirm the absence of an organic heart disease during follow up. Treatment of these benign arrhythmias doesn't required use of potent anti-arrhythmic drugs because of their potential side effects. However, the occurrence of this type of extrasystoles may generate concern in patients despite the assurances of the physician, and consequently worse quality of life. For these reasons it has been suggested treatment with a nutritional supplement, able to normalize the 'cardiac electrophysiology' and help to maintain wellness . Ritmonutra ® is a combination of nutraceuticals with a demonstrated efficacy on preserving the physiological cardiovascular functions in addition to an adequate diet. Ritmonutra ® is classified by the Ministry of Health as a food supplement with Notification in 26 Settmbre 2011. The functional components of Ritmonutra ®, including Omega-3 polyunsaturated fatty acids, Hawthorn, Astaxanthin and Vitamin E, help to normalize the pace, reducing the total number of benign extrasystoles, and consequently improving the quality of life. According to preliminary studies performed in patients with benign extrasystoles, both supraventricular and ventricular, free of specific heart disease, Ritmonutra ® has been demonstrated to have a significant effect in reducing the number of total extrasystoles and in improving the wellness of the subject. In particular, Ritmonutra ® was shown to improve the social life of individuals and reduce the limitations caused by emotional state, without side effects.
2. AIM OF THE STUDY

   Aim of the study is to investigate whether addition of Ritmonutra in addition to a adequate diet can improve and normalize the regular rhythm in patients free of specific organic cardiovascular disease compared to a mere placebo. Moreover, in patients with symptomatic benign extrasytoles, the investigators want to evaluate whether this nutraceutical supplement can reduce the discomfort related to perceiving these arrhythmias and consequently improve life quality.
3. STUDY DESIGN multicentre, randomized, controlled parallel-group study.
4. STUDY POPULATION The study will include participation of one clinic centre coordinating 150 general practitioners (GPs). Each GP will select at least 10 subjects of both gender, All participants will give written informed consent to the protocol approved by the local institutional review boards. At least 150 doctors will take part in the study; each will treat at least 10 subjects of both genders with diagnosis of symptomatic benign ventricular and supraventricular extrasytoles, free of specific organic cardiovascular disease and not requiring pharmacological therapy.

   Indicators:

   GPs are required: 1) to record a full medical history, including smoking and drinking habits, based on a pre-defined clinical record; 2) to collect demographic and anthropometric measures (height, weight, waist circumference at the iliac crest); 3) to perform a complete physical exam. At the first visit and after 4 and 8 weeks all eligible patients will perform a complete physical exam that includes measure of office blood pressure and heart rate in the sitting position and in triplicate, using a manual sphygmomanometer, according to international guidelines. Measurements will be rounded to the closest 2 mmHg interval. The baseline visit and the others screening visits also include Electrocardiogram (ECG), Ergometric test, Echocardiogram and Holter ECG.

   The primary endpoint is reduction of total number of extrasystoles. Secondary endpoint: the improvement in the wellness of the subject and consequently in the life quality.

   4.1. Sample size The estimate of the sample size was performed by the SISA method (Simple Interactive Statistical Analysis) - Machin, David and Campbell, Michael J. (1987) Statistical Tables for the Design of Clinical Trials. Blackwell Scientific Publications, Boston. Based on the values of a previous preliminary study comparing Ritmonutra ® with a control group (-58.5% reduction of total extrasystoles after 4 weeks with Ritmonutra ® compared with-0.5% in the control group) an approximate estimate was made of the number of observations necessary so that the two percentages are significant at the 5% probability level: 12 subjects cases in each group.
5. TREATMENTS

   All subjects will receive dietary counseling determined by the general practitioner depending on the subject's clinical condition, in accordance with the instructions of the Coordinating Site. Centralized randomization will be used to assign subjects to one of the two study treatments, Inert Placebo - Vitamin B complex + diet or vitamin B complex - Ritmonutra ® + diet. How Ritmonutra will be taken: 2 tavgel gum daily of Ritmonutra ® or vitamin B complex 2 tablets chewing a day.

   Duration of treatment: Subjects in both groups will take the assigned treatment for 4 weeks. Ritmonutra ® contains: 720 mg of Fish Oil with Omega-3, including 480 mg of EPA and 40 mg of DHA, Hawthorn (extract from Crataegus mongyna) 300 mg equivalent to 5.4 mg of vitexin, 4 mg of Astaxanthin and 36 mg of Vitamin E.
6. EVALUATION CRITERIA At baseline, and after 4 and 8 weeks cardiovascular parameters (blood pressure, heart rate, Holter ECG) and the SF-36 quality of life questionnaire and the 4SQ_2011questionnaire investigating somatic symptoms related to stress will be assessed as well as the others clinical parameters necessary to evaluate the cardiovascular risk and changes in life quality.
7. STUDY PROCEDURES Each doctor will initially be given a login and password allowing confidential and individual access to the website www.ritmonutra.net for data entry. In order to avoid sampling errors, the doctor will include in the study the first 10 consecutive subjects who meet the admission criteria (see point 4). The doctor will complete the appropriate form (also available on the ritmonutra.net site) insert information of the point 0 and will assign the subject to one of two regimens, Inert Placebo - Vitamin B complex + diet or vitamin B complex - Ritmonutra ® + diet, based on what has been determined by centralized randomization under the responsibility of Prof. Bruno Trimarco and delivery to the subject the treatment required for 4 weeks (Ritmonutra ® or control). After four weeks all the subjects under go to Holter ECG, the SF-36 and 4SQ_2011. After the first four weeks patients will receive the alternative treatment provided by randomization (control - Ritmonutra ®). After another four weeks all the subjects underwent 24-Hour Holter (ECG) monitoring , the SF-36 and 4SQ_2011.
8. STATISTICAL ANALYSIS The statistical analysis of baseline homogeneity will be undertaken using the chi-square test and analysis of variance, if appropriate.

   The statistical analysis to assess the clinical efficacy will be based on a comparison between differences at the various time points versus the baseline obtained in the two treatment groups and will be conducted using the chi-square test and analysis of variance, where appropriate.

   The level of significance will be considered to be an Alfa = 0.05 (type I error) and the power level a beta = 0.90 (type II error).
9. STUDY TIMELINES The study will start from the time the login and password have been delivered.
10. AVAILABILITY OF DATA All participants will be informed of the results once the data have been processed.
11. COORDINATING COMMITTEE

For any clarification on the study contact:

Dr. Claudio Benvenuti - Medical Management Rottapharm | Madaus Valosa via di Sopra, 9-20900 Monza tel 039 7390406 - Fax 039 7390393 email: @ claudio.benvenuti rottapharm.com.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ventricular or atrial extrasystoles

Exclusion Criteria:

* Presence of organic cardiomyopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction of the ventricular and atrial arrhythmias. | 4 week

SECONDARY OUTCOMES:
Improvement in life quality | 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, MD, Study Director — Federico II University, Dipartimento di medicina Clinica Scienze Cardiovascolari ed Immunologiche
Locations (1):
- Ambulatorio Ipertensione e Unità Coronarica Federico II University, Naples, Italy

REFERENCES:
- [Result] Izzo R, de Simone G, Giudice R, Chinali M, Trimarco V, De Luca N, Trimarco B. Effects of nutraceuticals on prevalence of metabolic syndrome and on calculated Framingham Risk Score in individuals with dyslipidemia. J Hypertens. 2010 Jul;28(7):1482-7. doi: 10.1097/HJH.0b013e3283395208. PMID 20498621
- See also: website of the High Blood Pressure Outpatient Clinic and UTIC of "Federico II" University of Naples — http://www.campaniasalute.com